CLINICAL TRIAL: NCT05723484
Title: A Multi-centre Diagnostic Study to Evaluate the Feasibility and Performance of the Genital InFlammation Test (GIFT)
Brief Title: Comparing a Novel Point-of-care Cytokine Biomarker Lateral Flow Test With Nucleic Acid Amplification Tests for Detection of Sexually Transmitted Infections and Bacterial Vaginosis
Acronym: GIFT
Status: Completed | Type: Observational
Sponsor: University of Cape Town (Other)
Collaborators: Macfarlane Burnet Institute for Medical Research and Public Health Ltd (Other); Desmond Tutu HIV Foundation (Other); London School of Hygiene and Tropical Medicine (Other); UMC Utrecht (Other); Institut Pasteur (Industry); Institut Pasteur de Madagascar (Other); Hitotsubashi University (Other)
Responsible Party: Principal Investigator, Jo-An Passmore, Professor, University of Cape Town
Other Study IDs: GIFT_EDCTP-RIA2020I-3297
Record Dates: First submitted 2023-01-27; First posted 2023-02-10 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-08

CONDITIONS: STI
MeSH Terms: conditions — Sexually Transmitted Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Urine - Pregnancy test Finger prick blood - HIV testing Dacron vaginal swab-SWAB 1 - GIFT device Dacron vaginal swab- SWAB 2 - Cytokine ELISA Dacron vaginal swab- SWAB 3 - pH Dacron vaginal swab-SWAB 3 - Nugent score Copan flocked vaginal swab- SWAB 4 - STI NAAT Copan flocked vaginal swab- SWAB 5 - STI NAAT Copan flocked vaginal swab- SWAB 5 - Quantitative PCR for Lactobacilli, Gardnerella vaginalis and Fannyhessea vaginae; Semen NAAT/ELISA Copan flocked vaginal swab-SWAB 6 and 7 - 16S rRNA sequencing
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Device: GIFT Device — The GIFT device - immune-based lateral flow test for reproductive-aged, non-pregnant in resource-limited settings attending sexual reproductive health (family planning) clinics, community health centers, hospitals, and mobile clinics. The test involves the qualitative detection of genital inflammation caused by asymptomatic STIs and BV in self- or clinician-collected lateral vaginal wall swabs, with results available in less than 20 minutes.

SUMMARY:
1. To evaluate the performance of a lateral flow POC test, namely the Genital InFlammation Test (GIFT), for identifying women with inflammatory STIs and BV, who are at higher risk of HIV infection and reproductive complications;
2. To evaluate how the GIFT device can be integrated in a feasible, acceptable, and cost-effective way into routine care.

DETAILED DESCRIPTION:
DIAGNOSTIC Study

Design:

The study is a multicentre, multidisciplinary, cross sectional, prospective clinically based research project.

The first component is a diagnostic study which will enrol 225 women attending family planning services in each of the three study sites in South Africa, Zimbabwe, and Madagascar. Vaginal samples from the women will be applied to the GIFT device and results will be compared with the composite NAAT reference test for STIs and Nugent score test for BV to determine the performance of the device to detect STIs/BV. Women will attend only one study visit but will be recalled for treatment if required.

The second component to develop a feasible, acceptable and economically feasible STI/BV management algorithm which includes the use of the GIFT device to be integrated into national guidelines (hereafter referred to as the "integration study") is composed of four activities with different study designs: 1.User experiences and/or perceptions of the GIFT device involving qualitative focus group discussions and in-depth interviews, and a quantitative questionnaire for health care professionals; 2. Discrete choice experiment; 3 Development of a decision tree classification algorithm; 4. Economic evaluation of the defined management algorithms.

Study Sites:

1. Cape Town, South Africa; Desmond Tutu Health Foundation (DTHF) Masiphumelele
2. Harare, Zimbabwe; Chitungwiza Primary Health Care Clinics
3. Antananarivo, Madagascar; Centre Hospitalier Universitaire Gynéco-Obstétrique de Befelatanana

Diagnostic Device:

The GIFT device is an immune-based lateral flow test for reproductive-aged, non-pregnant in resource-limited settings attending sexual reproductive health (family planning) clinics, community health centers, hospitals, and mobile clinics. The test involves the qualitative detection of genital inflammation caused by asymptomatic STIs and BV in self- or clinician-collected lateral vaginal wall swabs, with results available in less than 20 minutes.

Diagnostic Study Objectives:

Primary objectives To assess the sensitivity and specificity of the GIFT device at the point-of-care in non-pregnant sexually active women aged 18-35 years accessing family planning services in South Africa, Zimbabwe, and Madagascar.

Secondary objectives To assess the predictive values of the GIFT device at the point-of-care in non-pregnant sexually active women aged 18-35 years accessing family planning services in South Africa, Zimbabwe, and Madagascar; To assess the performance of the GIFT device at the point-of-care in non-pregnant sexually active women aged 18-35 years accessing family planning services in each of the countries; To assess the performance of the device versus syndromic management without any laboratory testing (standard of care in South Africa, Zimbabwe, and Madagascar); To determine the robustness of the device by comparing results read by clinicians with those read by laboratory professionals, and with the results obtained using an automated reader; To evaluate the accuracy of the GIFT device by comparing the GIFT device results with ELISA (enzyme-linked immunosorbent assay) results using previously validated concentration cut-offs as the gold standard, including validation of the GIFT cytokine concentration cut-offs for each cytokine biomarker.

Exploratory objectives Determine if other determinants (such as intermediate microbiota (Nugent 4-6), age, parity, sexual activity) improve the prediction of STI/BV status in women; To use 16S rRNA gene sequencing and vaginal bacteria specific quantitative NAATs to evaluate the proportion of cases of genital inflammation explained by vaginal dysbiosis that was not diagnosed as an STI or BV by NAATs or Nugent scoring; To explore the performance of the device in the presence of vaginal Candida spp colonisation.

INTEGRATION Study To evaluate how the GIFT device can be integrated in a feasible, acceptable, and cost-effective way into routine care (the "integration study"), four activities will be conducted: 1. User experiences and/or perceptions of the GIFT device; 2. Discrete choice experiment; 3 Development of a decision tree classification algorithm; 4. Economic evaluation of the defined management algorithms.

Objectives:

Primary objective To evaluate how the GIFT device could be integrated into routine care.

Secondary objectives To qualitatively and quantitatively assess the user-experience, usability, and acceptability of the GIFT device at the point of care; To examine patient preferences for various STI management aspects (attributes) to inform the development of STI management algorithms that integrate the GIFT device; To generate algorithms that integrate the GIFT device to optimise case finding and STIs/vaginal infection management in women, using the complete dataset from the study; To determine the cost and budget impact of the identified screening or diagnostic algorithm with the GIFT device, and to model the cost- effectiveness of different strategies of integration of GIFT into care.

ELIGIBILITY:
Diagnostic Inclusion Criteria:

* 18-35 years old
* Willing and able to provide informed consent to participate in the study
* Self-reported to be sexually active
* Not pregnant (determined by pregnancy test)
* Accessing family planning service

Integration Inclusion Criteria:

For all: Willing and able to provide informed consent to participate in the study

User experiences/perceptions activity:

* Local or regional policy makers, programmers and other opinion leaders and decision makers
* Healthcare professionals at health facilities
* Women who are eligible for the diagnostic study (including pregnant and menstruating women), but who are not part of the diagnostic study
* 18-35 years old
* Willing and able to provide informed consent to participate in the study
* Self-reported to be sexually active
* Accessing family planning service diagnostic study

Discrete choice experiments:

* Women who are eligible for the diagnostic study (including pregnant and menstruating women), who are either part of, or not part of, the diagnostic study
* 18-35 years old
* Self-reported to be sexually active
* Accessing family planning service diagnostic study

Decision tree classification algorithm:

* Data from diagnostic study participants

Economic evaluation:

* Healthcare professionals at health facilities involved in GIFT device implementation able to complete timesheets

Diagnostic Exclusion Criteria:

* <18 years or >35 years
* Refusal by a participant to participate in the study
* Treatment for any STI/BV in the past 30 days
* Pregnancy
* Enrolled in a study which does not allow co-enrolment in other studies

Integration Exclusion Criteria:

For all: Not willing or able to provide informed consent to participate in the study

User experiences/perceptions activity:

* Non-relevant policy makers
* Healthcare professionals at health facilities not included in diagnostic study

Women who are:

* Part of the diagnostic study
* <18 years or >35 years
* Treated for any STI/BV in the past 30 days
* Pregnant
* Enrolled in a study which does not allow co-enrolment in other studies

Discrete choice experiments:

Women who are:

* <18 years or >35 years
* Treated for any STI/BV in the past 30 days
* Pregnant
* Enrolled in a study which does not allow co-enrolment in other studies

Decision tree classification algorithm:

* Participants for whom there are no diagnostic study data

Economic evaluation:

* Healthcare professionals not at study sites, not involved in GIFT device implementation, and/or not able to complete timesheets

Ages: 18 Years to 35 Years | Sex: Female
Age Groups: Adult
Study Population: Diagnostic:
  Non-pregnant, sexually active women aged 18-35 years accessing family planning services.
  Integration:
  * Local or regional policy makers: maximum 36
  * Healthcare professionals: maximum 40
  * Pregnant and non-pregnant, sexually active women of 18-35 years attending family planning services: maximum 45
  * Pregnant and non-pregnant, sexually active women of 18-35 years attending family planning services: up to 200 participants per site for discrete choice experiment
  * Data from pregnant and non-pregnant, sexually active women of 18-35 years attending family planning services recruited in diagnostic study
  * Healthcare workers from diagnostic study sites
Sampling Method: Probability Sample
Enrollment: 675 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Estimates of sensitivity and specificity for the GIFT device | Start- quarter 1/2023; End- quarter 4/2023
  Detecting the presence of any STI or BV with 95% confidence intervals, using NAATs and Nugent scoring in a composite reference standard.
How the GIFT device could be integrated into routine care | Start- quarter 1/2023; End- quarter 4/2023
  Integration into healthcare guidelines

SECONDARY OUTCOMES:
Positive and negative predictive values of the GIFT device | Start- quarter 1/2023; End- quarter 4/2023
  predictive values of the GIFT device in each country and likelihood ratios, using NAATs and Nugent scoring as a composite reference standard
Overall sensitivity of NAAT and Nugent scoring | Start- quarter 1/2023; End- quarter 4/2023
  Specificity and predictive values in each country using NAATs and Nugent scoring
Overall sensitivity | Start- quarter 1/2023; End- quarter 4/2023
  Specificity and predictive values in each country and likelihood ratios of syndromic management, using NAATs and Nugent scoring as composite reference standards
Comparison of sensitivity, specificity, predictive values in each country and likelihood ratios calculated with both methods | Start- quarter 1/2023; End- quarter 4/2023
  GIFT device and syndromic management using NAATs and Nugent scoring as composite reference standards
Positive and negative agreement proportion and Kappa coefficient between results readings of 1/clinician and technician | Start- quarter 1/2023; End- quarter 4/2023
  2/clinician and automated reader; 3/technician and automated reader
Positive and negative agreement proportion and Kappa coefficient between results readings of GIFT device and cytokine ELISA measurements | Start- quarter 1/2023; End- quarter 4/2023
  GIFT device and cytokine ELISA measurements
User experiences | Start- quarter 1/2023; End- quarter 4/2023
  Perceptions of GIFT device
User preferences | Start- quarter 2/2023; End- quarter 1/2024
  different STI management strategies based on patient preferences for various attributes of STI management using GIFT device
Optimal case finding and STI management strategies | Start: - quarter 1/2024; End- quarter 4/2024
  Using diagnostic study results
Cost and budget impact | Start- quarter 3/2023; End- quarter 2/2024
  Economic evaluation for the budget impact analysis to create strategies of integrating the GIFT device into standard of care

OTHER OUTCOMES:
Expository Endpoint: Post-estimation classifications | Start- quarter 3/2023; End- quarter 4/2024
  (% of women correctly classified, fit of the model) from logistic regression models.

CONTACTS AND LOCATIONS:
Overall Officials: Jo-Ann Passmore, Professor, Principal Investigator — University of Cape Town
Locations (3):
- Centre Hospitalier Universitaire Gynéco-Obstétrique de Befelatanana, Antananarivo, Madagascar
- Desmond Tutu Health Foundation, Cape Town, Western Cape, South Africa
- Chitungwiza Primary Health Care Clinics, Harare, Zimbabwe

IPD SHARING:
Plan to Share IPD: No
De-identified study data will be made available to the study team only.

REFERENCES:
- [Derived] Ramboarina S, Crucitti T, Gill K, Bekker LG, Harding-Esch EM, van de Wijgert JHHM, Huynh BT, Fortas C, Harimanana A, Mayouya Gamana T, Randremanana RV, Mangahasimbola R, Dziva Chikwari C, Kranzer K, Mackworth-Young CRS, Bernays S, Thomas N, Anderson D, Tanko FR, Manhanzva M, Lurie M, Khumalo F, Sinanovic E, Honda A, Pidwell T, Francis SC, Masson L, Passmore JA; GIFT study group. Novel point-of-care cytokine biomarker lateral flow test for the screening for sexually transmitted infections and bacterial vaginosis: study protocol of a multicentre multidisciplinary prospective observational clinical study to evaluate the performance and feasibility of the Genital InFlammation Test (GIFT). BMJ Open. 2024 May 1;14(5):e084918. doi: 10.1136/bmjopen-2024-084918. PMID 38692732